CLINICAL TRIAL: NCT03642990
Title: Nicotinamide Riboside (NR) in Paclitaxel-induced Peripheral Neuropathy
Brief Title: NR in Chemo-induced Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment challenges
Sponsor: Donna Hammond, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH); ChromaDex, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Donna Hammond, PhD, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201612723; R21CA208968 (NIH)
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Breast Cancer Metastatic; Platinum-resistant Recurrent Ovarian Cancer; Head and Neck Cancer Stage IV; Endometrial Cancer Stage IV
Keywords: paclitaxel; nicotinamide riboside; NIAGEN; nab-paclitaxel
MeSH Terms: conditions — Head and Neck Neoplasms; Endometrial Neoplasms | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: All subjects with stage IV breast cancer, platinum-resistant recurrent ovarian, peritoneal, endometrial, or fallopian tube cancer, or platinum-resistant recurrent or metastatic head and neck cancer will receive 300 mg NIAGEN®) daily for one week followed by dose escalation to 1000 mg daily for 11 weeks upon reporting the development of grade 1 sensory neuropathy. Those presenting with a residual sensory neuropathy of ≤ 2 as a result of prior chemotherapy will also be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NIAGEN®) (Experimental): Daily oral administration of nicotinamide riboside 300 mg (150 mg a.m. and p.m.) for one week with dose escalation to 1000 mg (500 mg a.m. and p.m.) for remaining 11 weeks.
  Interventions: Drug: Nicotinamide Riboside

INTERVENTIONS:
Drug: Nicotinamide Riboside — Capsule
  Other Names: NIAGEN®)

SUMMARY:
The purpose of this single-arm phase II trial is to determine whether nicotinamide riboside (NIAGEN®) prevents the progression of peripheral sensory neuropathy in patients receiving infusions of paclitaxel or nab-paclitaxel for the treatment of metastatic breast cancer or recurrent platinum-resistant ovarian, endometrial, peritoneal, fallopian tube cancer or metastatic head and neck cancer.

DETAILED DESCRIPTION:
Peripheral neuropathies are a dose-limiting, disabling, and debilitating side effect of virtually every known class of chemotherapeutic agent, and are referred to as chemotherapy-induced peripheral neuropathies (CIPN) (Seretny et al., 2014). The incidence and severity of CIPN increase as the cumulative dose, frequency of administration, and the number of therapeutic cycles increase. As many as 68% of patients have CIPN when assessed within 30 days of completing treatment. Patients experience paresthesias, dysesthesias (an unpleasant abnormal sensation, whether spontaneous or evoked), hyperalgesia (increased pain from a stimulus that normally provokes pain), allodynia (pain due to a stimulus that does not normally provoke pain), numbness or loss of sensation, or ongoing pain that is burning, lancinating or electric shock-like in nature. CIPN can seriously diminish a patient's quality of life, and can interfere with self-care and activities of daily living. The severity of CIPN may also necessitate reducing the dose of chemotherapeutic agent, delaying the next cycle of chemotherapy, or terminating treatment entirely (Argyriou et al., 2012; Argyriou et al., 2014; Miltenburg et al., 2014; Park et al., 2013).

Nicotinamide adenine dinucleotide (NAD+) is an essential redox coenzyme required for cell viability, basic bioenergetics, and fast axonal transport (Yang and Sauve, 2016). It plays an important role in protection against axonal injury from either mechanical or neurotoxic injury (Araki et al., 2004; Sasaki et al., 2006; Sasaki et al., 2009; Gerdts et al., 2015; Khan et al., 2014; Conforti et al., 2014; Di Stefano et al., 2015). Nicotinamide riboside (NIAGEN®) is a form of vitamin B3 and a precursor in the pathway for synthesis of NAD+ (Bieganowski et al., 2004; Trammell et al., 2016; Chi and Sauve, 2013). Oral administration of NIAGEN® increases levels of NAD+ in the blood, liver, skeletal muscle, and other tissues (Canto et al., 2012; Hamity et al, 2017; Airhart et al., 2017; Martens et al., 2018).

NIAGEN®) has been reported to prevent tactile hypersensitivity and blunt the affective dimension of nociception in a rat model of CIPN (Hamity et al., 2017) It also prevents signs of peripheral neuropathy in a mouse model of diabetes (Trammell et al., 2016) The proposed single-arm pilot phase II study will examine whether daily dosing with NIAGEN®) can prevent the progression of CIPN in persons with stage IV breast cancer or recurrent platinum-resistant ovarian, endometrial, peritoneal, or fallopian tube cancer receiving once weekly infusions of paclitaxel for 12 weeks.

In this study, persons with metastatic breast cancer, platinum-resistant recurrent ovarian, peritoneal, endometrial, or fallopian tube cancer, or platinum-resistant recurrent or metastatic head and neck cancer who are receiving weekly infusions of paclitaxel or nab-paclitaxel and anticipated to survive for at least 3 months will be offered the opportunity to enroll in this study when they develop a peripheral neuropathy of at least grade 1. Persons with peripheral neuropathy of no greater than a grade 2 from prior therapy may also enroll in this study if they are receiving weekly infusions of paclitaxel or nab-paclitaxel. Upon enrollment, health care providers will review the overall severity of the participant's neuropathy and assign a baseline grade. Participants will also complete two short questionnaires that will more specifically score how the peripheral neuropathy interferes with daily functions of living. A small sample of blood will be taken at the completion of the paclitaxel or nab-paclitaxel infusion to measure levels of paclitaxel. The participant will then be sent home with capsules of NIAGEN® to take twice daily. Each week upon return to the clinic a small sample of blood will be taken before the infusion of paclitaxel to measure biomarkers for NIAGEN®, and other samples of blood will be taken to evaluate clinical chemistries, kidney, and liver function. Another sample of blood will be obtained after the paclitaxel or nab-paclitaxel infusion to measure levels of paclitaxel or nab-paclitaxel. The health care provider will meet with the patient each week to score the overall severity of the peripheral neuropathy, and the participant will answer another questionnaire with more specific questions. Once a month, the participant will be asked to fill out a second questionnaire. Participants will take 300 mg/day NIAGEN® in the first week and 1000 mg/day in the subsequent 11 weeks. The study will conclude one week after the 12th infusion of paclitaxel or nab-paclitaxel. Health care providers will contact the participant at various times up to 6 months to monitor their status.

Beginning with completion of the trial by the 10th participant and continuing with each subsequent participant up to 39, we will use a Bayesian statistical approach (Lee and Liu, 2008; i.e. predictive probability) to determine whether NIAGEN® has prevented a worsening of the peripheral neuropathy. This approach we let us make an early determination of futility. We will also determine whether NIAGEN® has decreased the need to delay or diminish the doses of paclitaxel or nab-paclitaxel due to severity of the peripheral neuropathy. The results of this trial will inform the design of a subsequent randomized, placebo-controlled, blinded clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent and HIPAA authorization
* Be 18 to 85 years old
* Have been diagnosed with stage IV breast cancer of any type, platinum-resistant recurrent ovarian, peritoneal, endometrial, or fallopian tube cancer, or platinum-resistant recurrent or metastatic head and neck cancer and are anticipated to survive for at least three months
* Have an ECOG Performance Status of 0-2
* Able to take medication orally - up to four capsules in the morning (am) and four capsules in the evening (pm).
* Be undergoing infusions of paclitaxel or nab-paclitaxel for treatment of breast cancer, platinum-resistant recurrent ovarian, peritoneal, endometrial, or fallopian tube cancer, or platinum-resistant recurrent or metastatic head and neck cancer and be determined to have at least a grade 1 neuropathy based on the CTCAE version 4.03 guidelines for peripheral sensory neuropathy. Breast cancer patients may also be treated concomitantly with monoclonal antibodies to HER2 such as trastuzumab (Herceptin) and pertuzumab (Perjeta). Patients with platinum-resistant ovarian, peritoneal, endometrial, or fallopian tube cancer or platinum-resistant recurrent or metastatic head and neck cancer may also be treated concomitantly with a vascular endothelial growth receptor 2 inhibitor such as bevacizumab (Avastin) or a checkpoint inhibitor.
* Females must be either postmenopausal for at least 1 year or surgically sterile for at least 6 weeks. Females of childbearing potential must have a negative pregnancy test at screening to be eligible for study participation, and agree to take appropriate precautions to avoid pregnancy from screening through follow-up.
* Males must agree to take appropriate precautions to avoid fathering a child from screening through follow-up. The following methods have been determined to be more than 99% effective (<1% failure rate per year when used consistently and correctly) and are permitted under this protocol for use by the patient and his/her partner:

  * Complete abstinence from sexual intercourse when this is in line with the preferred and usual lifestyle of the patient
  * Double barrier methods including condom with spermicide in conjunction with use of an intrauterine device or condom with spermicide in conjunction with use of a diaphragm
* Surgical sterilization (bilateral oopherectomy with or without hysterectomy, tubal ligation or vasectomy) at least 6 weeks prior to taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up levels of luteinizing hormone (LH), follicle-stimulating hormone (FSH), and/or estradiol.

Non-hormonal intrauterine device used as directed by provider placing this is also acceptable.

Exclusion Criteria:

* Pre-existent peripheral neuropathy that is unrelated to chemotherapy
* Pre-existent chemotherapy-induced peripheral neuropathy greater than grade 2
* Known metastases to the brain, spinal cord or peripheral nerves, or leptomeningeal disease
* Concurrent administration of a poly (ADP-Ribose) polymerase inhibitor (e.g. olaparib, rucaparib)
* Concurrent administration of a platinum-based chemotherapy
* Diabetes requiring management by medication
* Diabetes managed by medication
* Neutrophils < 1,000 cells/m3
* Hemoglobin < 8.0 g/dcl
* Platelets < 100,000 cells/m3
* Creatinine clearance < 30 ml/min
* AST or ALT values > 2.5 X upper limits of normal
* Total bilirubin > 2.0 X upper limits of normal
* Heavy alcohol use defined at > 8 drinks/week by women or 12 drinks/week by men
* Chronic pain greater than 3 months duration within the past year.
* Severe psychiatric illness
* Pregnancy
* Current imprisonment
* Limitations of self-expression, defined as an inability to answer questions posed by physicians, nurses, care-givers, or other members of the investigative team or an inability to describe somatosensations.
* Known HIV, not on therapy
* Regular use of nutritional supplements that contain nicotinamide or NIAGEN® within the previous 30 days
* Use of duloxetine (Cymbalta®) within the previous 30 days
* Pancreatic insufficiency requiring exocrine enzyme replacement therapy
* GI conditions where malabsorption of B complex vitamins is known to occur.
* Known allergy to Cremophor vehicle used to deliver paclitaxel in its Taxol formulation
* Breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2022-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna L Hammond, PhD, Principal Investigator — University of Iowa; Alexandra Thomas, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification, will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. The IPD will be available to sharing immediately after publication and ending 5 years after article publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years after article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.

REFERENCES:
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Argyriou AA, Bruna J, Marmiroli P, Cavaletti G. Chemotherapy-induced peripheral neurotoxicity (CIPN): an update. Crit Rev Oncol Hematol. 2012 Apr;82(1):51-77. doi: 10.1016/j.critrevonc.2011.04.012. Epub 2011 Sep 10. PMID 21908200
- [Background] Argyriou AA, Kyritsis AP, Makatsoris T, Kalofonos HP. Chemotherapy-induced peripheral neuropathy in adults: a comprehensive update of the literature. Cancer Manag Res. 2014 Mar 19;6:135-47. doi: 10.2147/CMAR.S44261. eCollection 2014. PMID 24672257
- [Background] Miltenburg NC, Boogerd W. Chemotherapy-induced neuropathy: A comprehensive survey. Cancer Treat Rev. 2014 Aug;40(7):872-82. doi: 10.1016/j.ctrv.2014.04.004. Epub 2014 Apr 18. PMID 24830939
- [Background] Park SB, Goldstein D, Krishnan AV, Lin CS, Friedlander ML, Cassidy J, Koltzenburg M, Kiernan MC. Chemotherapy-induced peripheral neurotoxicity: a critical analysis. CA Cancer J Clin. 2013 Nov-Dec;63(6):419-37. doi: 10.3322/caac.21204. PMID 24590861
- [Background] Bieganowski P, Brenner C. Discoveries of nicotinamide riboside as a nutrient and conserved NRK genes establish a Preiss-Handler independent route to NAD+ in fungi and humans. Cell. 2004 May 14;117(4):495-502. doi: 10.1016/s0092-8674(04)00416-7. PMID 15137942
- [Background] Trammell SA, Yu L, Redpath P, Migaud ME, Brenner C. Nicotinamide Riboside Is a Major NAD+ Precursor Vitamin in Cow Milk. J Nutr. 2016 May;146(5):957-63. doi: 10.3945/jn.116.230078. Epub 2016 Apr 6. PMID 27052539
- [Background] Chi Y, Sauve AA. Nicotinamide riboside, a trace nutrient in foods, is a vitamin B3 with effects on energy metabolism and neuroprotection. Curr Opin Clin Nutr Metab Care. 2013 Nov;16(6):657-61. doi: 10.1097/MCO.0b013e32836510c0. PMID 24071780
- [Background] Hamity MV, White SR, Walder RY, Schmidt MS, Brenner C, Hammond DL. Nicotinamide riboside, a form of vitamin B3 and NAD+ precursor, relieves the nociceptive and aversive dimensions of paclitaxel-induced peripheral neuropathy in female rats. Pain. 2017 May;158(5):962-972. doi: 10.1097/j.pain.0000000000000862. PMID 28346814
- [Background] Trammell SA, Weidemann BJ, Chadda A, Yorek MS, Holmes A, Coppey LJ, Obrosov A, Kardon RH, Yorek MA, Brenner C. Nicotinamide Riboside Opposes Type 2 Diabetes and Neuropathy in Mice. Sci Rep. 2016 May 27;6:26933. doi: 10.1038/srep26933. PMID 27230286
- [Background] Lee JJ, Liu DD. A predictive probability design for phase II cancer clinical trials. Clin Trials. 2008;5(2):93-106. doi: 10.1177/1740774508089279. PMID 18375647
- [Background] Yang Y, Sauve AA. NAD(+) metabolism: Bioenergetics, signaling and manipulation for therapy. Biochim Biophys Acta. 2016 Dec;1864(12):1787-1800. doi: 10.1016/j.bbapap.2016.06.014. Epub 2016 Jun 29. PMID 27374990
- [Background] Araki T, Sasaki Y, Milbrandt J. Increased nuclear NAD biosynthesis and SIRT1 activation prevent axonal degeneration. Science. 2004 Aug 13;305(5686):1010-3. doi: 10.1126/science.1098014. PMID 15310905
- [Background] Sasaki Y, Araki T, Milbrandt J. Stimulation of nicotinamide adenine dinucleotide biosynthetic pathways delays axonal degeneration after axotomy. J Neurosci. 2006 Aug 16;26(33):8484-91. doi: 10.1523/JNEUROSCI.2320-06.2006. PMID 16914673
- [Background] Sasaki Y, Vohra BP, Lund FE, Milbrandt J. Nicotinamide mononucleotide adenylyl transferase-mediated axonal protection requires enzymatic activity but not increased levels of neuronal nicotinamide adenine dinucleotide. J Neurosci. 2009 Apr 29;29(17):5525-35. doi: 10.1523/JNEUROSCI.5469-08.2009. PMID 19403820
- [Background] Sasaki Y, Vohra BP, Baloh RH, Milbrandt J. Transgenic mice expressing the Nmnat1 protein manifest robust delay in axonal degeneration in vivo. J Neurosci. 2009 May 20;29(20):6526-34. doi: 10.1523/JNEUROSCI.1429-09.2009. PMID 19458223
- [Background] Gerdts J, Brace EJ, Sasaki Y, DiAntonio A, Milbrandt J. SARM1 activation triggers axon degeneration locally via NAD(+) destruction. Science. 2015 Apr 24;348(6233):453-7. doi: 10.1126/science.1258366. Epub 2015 Apr 23. PMID 25908823
- [Background] Khan NA, Auranen M, Paetau I, Pirinen E, Euro L, Forsstrom S, Pasila L, Velagapudi V, Carroll CJ, Auwerx J, Suomalainen A. Effective treatment of mitochondrial myopathy by nicotinamide riboside, a vitamin B3. EMBO Mol Med. 2014 Jun;6(6):721-31. doi: 10.1002/emmm.201403943. PMID 24711540
- [Background] Conforti L, Gilley J, Coleman MP. Wallerian degeneration: an emerging axon death pathway linking injury and disease. Nat Rev Neurosci. 2014 Jun;15(6):394-409. doi: 10.1038/nrn3680. PMID 24840802
- [Background] Di Stefano M, Nascimento-Ferreira I, Orsomando G, Mori V, Gilley J, Brown R, Janeckova L, Vargas ME, Worrell LA, Loreto A, Tickle J, Patrick J, Webster JR, Marangoni M, Carpi FM, Pucciarelli S, Rossi F, Meng W, Sagasti A, Ribchester RR, Magni G, Coleman MP, Conforti L. A rise in NAD precursor nicotinamide mononucleotide (NMN) after injury promotes axon degeneration. Cell Death Differ. 2015 May;22(5):731-42. doi: 10.1038/cdd.2014.164. Epub 2014 Oct 17. PMID 25323584
- [Background] Martens CR, Denman BA, Mazzo MR, Armstrong ML, Reisdorph N, McQueen MB, Chonchol M, Seals DR. Chronic nicotinamide riboside supplementation is well-tolerated and elevates NAD+ in healthy middle-aged and older adults. Nat Commun. 2018 Mar 29;9(1):1286. doi: 10.1038/s41467-018-03421-7. PMID 29599478
- [Background] Airhart SE, Shireman LM, Risler LJ, Anderson GD, Nagana Gowda GA, Raftery D, Tian R, Shen DD, O'Brien KD. An open-label, non-randomized study of the pharmacokinetics of the nutritional supplement nicotinamide riboside (NR) and its effects on blood NAD+ levels in healthy volunteers. PLoS One. 2017 Dec 6;12(12):e0186459. doi: 10.1371/journal.pone.0186459. eCollection 2017. PMID 29211728
- [Background] Canto C, Houtkooper RH, Pirinen E, Youn DY, Oosterveer MH, Cen Y, Fernandez-Marcos PJ, Yamamoto H, Andreux PA, Cettour-Rose P, Gademann K, Rinsch C, Schoonjans K, Sauve AA, Auwerx J. The NAD(+) precursor nicotinamide riboside enhances oxidative metabolism and protects against high-fat diet-induced obesity. Cell Metab. 2012 Jun 6;15(6):838-47. doi: 10.1016/j.cmet.2012.04.022. PMID 22682224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were approached at two sites: University of Iowa and Wake Forest Baptist Medical Center. All five subjects enrolled in the study were at Wake Forest Baptist Medical Center.
Pre-assignment Details: Seven subjects were screened for enrollment, of whom two were ineligible.
Period: 300 mg/Day for One Week
Arm/Group | NIAGEN®)
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: 1000 mg/Day for Weeks 2-12
Arm/Group | NIAGEN®)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | NIAGEN®)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
NAD concentration plasma levels [Mean (Inter-Quartile Range); unit: micrograms/ml] — Plasma sample obtained before NIAGEN treatment begun
  micrograms/ml | 27.5 [25.9 to 50.3]
1-methyl-nicotinamide plasma levels [Median (Inter-Quartile Range); unit: ng/ml] — Plasma samples obtained before NIAGEN treatment begun
  ng/ml | 11.1 [6.35 to 187]
paclitaxel plasma levels [Median (Inter-Quartile Range); unit: ng/ml] — Plasma sample obtained 10-20 min after taxane infusion ended Population: one sample not submitted due to subject testing COVID positive and withdrawing from study
  ng/ml
    number analyzed (Participants) | 4
    (all) | 1629 [1019 to 2564]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With No Worsening in the Grade of Peripheral Sensory Neuropathy as Scored by CTCAE
Description: The primary outcome variable is defined as no worsening of the grade of peripheral sensory neuropathy as scored according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 guidelines. Per the CTCAE a score of 1 would be assigned in the instance of parethesias or a loss of deep tendon reflexes. A score of 2 would be assigned in the instance of moderate symptoms that limit instrumental activities of daily living. A score of 3 would be assigned in the instance of severe symptoms that limit self-care activities of daily living. Because the outcome measure is defined as no worsening of the grade, it was recorded as either "yes"( i.e. it worsened) or "no" (i.e. it did not worsen).
Time Frame: approximately 4 weeks
Population: Data are reported for the 4 subjects who took at least one dose of NIAGEN. End of treatment was originally defined as within 2 weeks after 12 weeks of NIAGEN treatment ended (i.e. a study duration of ~14 weeks). If a patient withdrew before completing 12 weeks of treatment, the end of treatment was designated as one week after withdrawal from the study. The longest that any participant was on NIAGEN was three weeks. Therefore, the time frame of the study has been adjusted to ~4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | NIAGEN®)
Number analyzed (Participants) | 4
Participants | 3

2. Secondary Outcome: Percentage of Patients in Which Dose of Paclitaxel or Nab-Paclitaxel is Reduced Due to CIPN
Description: Quantitate the percentage of patients that experience a dose reduction of paclitaxel or nab-paclitaxel therapy due to neuropathy.
Time Frame: 3 weeks
Population: Data are reported for the only subject who received more than 1 dose of taxane chemotherapy before withdrawal from the trial. That subject patient received only 2 doses of taxane over a period of 3 weeks. No patient completed the full 12 weeks of the trial. Therefore, the time frame of the study has been adjusted from the originally envisioned 12 weeks to ~3 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | NIAGEN®)
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Number of Dose Reduction Events
Description: Count the number of (i.e. the incidence) of dose reduction events due to neuropathy (each occasion of dose reduction is a separate event);
Time Frame: 3 weeks
Population: Data are reported for the only subject who received more than 1 dose of taxane chemotherapy before withdrawal from the trial. That patient received only 2 doses of taxane over a period of 3 weeks. The original aim was to assess dose reduction over the 12 weeks of paclitaxel treatment, but no patient completed the 12 weeks of treatment. As the longest that any patient was on NIAGEN was 3 weeks, the time frame has been adjusted accordingly.
Measure: Number; unit: event
Arm/Group | NIAGEN®)
Number analyzed (Participants) | 1
event | 0

4. Secondary Outcome: Total Dose of Paclitaxel Administered
Description: Quantitate the total cumulative dose of paclitaxel administered over the 12 weeks.
Time Frame: 3 weeks
Population: Data are reported for the 1 subject who received taxane infusions after starting NIAGEN treatment. They received 2 infusions over a period of three weeks of NIAGEN treatment.
Measure: Number; unit: mg/M^2
Arm/Group | NIAGEN®)
Number analyzed (Participants) | 1
mg/M^2 | 200

5. Secondary Outcome: Difference in Score Between Baseline and End of Treatment for the FACT&GOG-NTX Subscale .
Description: Difference in Score on the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - neurotoxicity questionnaire at the end of treatment; i.e. Score at screening - score at end of treatment. This questionnaire asks 11 questions that are specific to chemotherapy-induced peripheral neuropathies. Maximum score is 44, minimum score is 0. Positive differences indicate a decrease in neuropathy. Negative differences indicate a worsening of neuropathy. Zero means unchanged.
Time Frame: 4 weeks
Population: Data are reported for the three subjects who took at least one dose of NIAGEN and completed the FACT questionnaire. End of treatment was originally defined as within 2 weeks after 12 weeks of NIAGEN treatment ended (i.e. a study duration of ~ 14 weeks). If a patient withdrew before then, the end of treatment was designated as one week after withdrawal. Unfortunately, the longest that any patient was on NIAGEN was three weeks. Therefore, the time frame has been adjusted to ~4 weeks.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | NIAGEN®)
Number analyzed (Participants) | 3
units on a scale | 7 [2 to 11]

6. Other Pre Specified Outcome: Difference in Total Neuropathy Score Between Screening and End of Treatment
Description: Exploratory analysis of ability of the clinical version of the Total Neuropathy Score questionnaire to detect changes in CIPN severity over time. Unlike the CTCAE or the FACT&GOG-NTX questionnaires, the TNS is a patient reported outcome measure. HIghest score (worse neuropathy is 24, lowest score is 0. Outcome assessed difference between end of treatment and screening. A positive number indicates improvement in neuropathy
Time Frame: 4 weeks
Population: Data are reported for the three subjects who took at least one dose of NIAGEN and completed the TNS evaluation. No patient completed the full 12 weeks of the trial. Therefore, the measure was made at end of treatment, which was designated as one week after they ceased NIAGEN treatment. The longest any one patient was on NIAGEN was three weeks. Hence the time frame was adjusted to 4 weeks.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | NIAGEN®)
Number analyzed (Participants) | 3
score on a scale | 2 [0 to 5]

7. Post Hoc Outcome: Plasma Concentration of Paclitaxel After NIAGEN Treatment Began
Description: Paclitaxel levels in plasma were measured ~30 min after each infusion of taxane. This was undertaken to ascertain whether NIAGEN altered plasma levels of paclitaxel because increases or decreases in plasma levels of paclitaxel by itself could lead to an apparent worsening or improvement, respectively, in CIPN and confound interpretation of NIAGEN's effect.
Time Frame: up to 3 weeks
Population: Data are reported for three subjects in which paclitaxel levels were obtained before NIAGEN and after NIAGEN treatment, which ranged from one to three weeks. The plasma concentration for the last blood sample obtained after NIAGEN treatment
Measure: Median (Full Range); unit: ng/ml
Arm/Group | NIAGEN®)
Number analyzed (Participants) | 3
ng/ml | 810 [259.7 to 1525]

ADVERSE EVENTS:
Time Frame: Up to six months after end of treatment (typically 7 months total)
Description: Subjects were queried for adverse events by phone interview 1, 3 and 6 months after end of treatment.
Arm/Group | NIAGEN®)
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIAGEN®) (N=5)
Nausea (Gastrointestinal disorders) | 4 (5)
mucositis oral (Gastrointestinal disorders) | 1 (2) — worsening pain from lesion
diarrhea (Gastrointestinal disorders) | 3 (3)
dyspepsia (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
headache (Nervous system disorders) | 3 (3)
peripheral sensory neuropathy (Nervous system disorders) | 2 (5)
dizziness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
peripheral motor neuropathy (Nervous system disorders) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
localized edema (General disorders) | 1 (1)
pain (General disorders) | 1 (1)
white blood cell decreased (Investigations) | 2 (4)
alanine aminotransferase increased (Investigations) | 1 (1)
lymphocyte count decreased (Investigations) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
chest pain (Cardiac disorders) | 1 (1)
upper respiratory infection (Infections and infestations) | 1 (3)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
flushing (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was limited to a non-curative population of women receiving taxane chemotherapy without added platinum-based agents. Difficulty in recruiting this small population led to eventual termination of the trial. Dose escalation to 1000 mg/day did not occur for any subject due to physician concerns that subjects were not tolerating the 300 mg dose well.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT03642990/Prot_SAP_003.pdf
  • Informed Consent Form: University of Iowa (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03642990/ICF_004.pdf
  • Informed Consent Form: Wake Forest (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03642990/ICF_005.pdf